CLINICAL TRIAL: NCT04683406
Title: A Randomized, Double-blind Phase III Clinical Study of ZSP1273 Tablets Compared With Placebo or Oseltamivir Patients With Acute Uncomplicated Influenza A
Brief Title: A Study of ZSP1273 Tablets in Patients With Acute Uncomplicated Influenza A
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guangdong Raynovent Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZSP1273-20-06
Record Dates: First submitted 2020-12-13; First posted 2020-12-24 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Influenza A
MeSH Terms: interventions — ZSP1273

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ZSP1273 600 mg + Oseltamivir Placebo BID (Experimental): Subjects received 5 doses of ZSP1273 at 600 mg once a day along with matching placebo of oseltamivir placebo orally twice daily (BID) with approximately 12 hour (+/- 2) intervals, over 5 days
  Interventions: Drug: ZSP1273 600 mg; Drug: Placebo to Oseltamivir
- Oseltamivir 75mg + ZSP1273 Placebo (Active Comparator): Subjects received 10 doses of Oseltamivir at a dose of 75 mg twice daily (BID) with matching placebo of ZSP1273 orally once a day with approximately 12 hour (+/- 2) intervals, over 5 days
  Interventions: Drug: Oseltamivir(oral); Drug: Placebo to ZSP1273
- Placebo Comparator (Placebo Comparator): Subjects received 5 doses of matching placebo of ZSP1273 and Oseltamivir twice daily (BID) with approximately 12 hour (+/- 2) intervals, over 5 days
  Interventions: Drug: Placebo to Oseltamivir; Drug: Placebo to ZSP1273

INTERVENTIONS:
Drug: ZSP1273 600 mg — 3 X 200-mg tablet taken orally
  Arms: ZSP1273 600 mg + Oseltamivir Placebo BID
Drug: Placebo to Oseltamivir — Placebo capsules matching oseltamivir2 X 75-mg
  Arms: Placebo Comparator; ZSP1273 600 mg + Oseltamivir Placebo BID
Drug: Oseltamivir(oral) — 2 X 75-mg tablet taken orally
  Arms: Oseltamivir 75mg + ZSP1273 Placebo
Drug: Placebo to ZSP1273 — Placebo capsules matching ZSP1273 600 mg
  Arms: Oseltamivir 75mg + ZSP1273 Placebo; Placebo Comparator

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled, and active controlled clinical trial to assess the efficacy and safety of ZSP1273 tablets in the treatment of Acute Uncomplicated influenza A.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are able to understand the study and comply with all study procedures, and willing to provide written informed consent/assent prior to the predose examinations appropriately.
2. Male or female patient s aged ≥ 18 to ≤ 64 years at the time of signing the informed consent/assent form
3. Patients with a diagnosis of influenza virus infection confirmed by all of the following

   * Positive Rapid Antigen Test (RAT) with throat swabs;and
   * Fever ≥ 38ºC (axillary) in the predose examinations or > 4 hours after dosing of antipyretics if they were taken;and
   * At least one of the following general systemic symptoms associated with influenza are present with a severity of moderate or greater I. Headache II. Feverishness or chills III. Muscle or joint pain IV. Fatigue
   * At least one of the following respiratory symptoms associated with influenza are present with a severity of moderate or greater I. Cough II. Sore throat III. Nasal congestion
4. The time interval between the onset of symptoms and the predose examinations is 48 hours or less. The onset of symptoms is defined as either

   * Time of the first increase in body temperature (an increase of at least 1ºC from normal body temperature)
   * Time when the patient experiences at least one general or respiratory symptom
5. Women of childbearing potential (WOCBP) who agree to use a highly effective method of contraception for 3 months after the first dose of ZSP1273 or oseltamivir

Exclusion Criteria:

1. Patients with severe influenza virus infection requiring inpatient treatment
2. Patients aged ≥ 18 years with known allergy to oseltamivir (Tamiflu) or ZSP1273
3. Patients unable to swallow tablets or capsules or any medical history in gastrointestinal that interferes with the absorption of drugs
4. Patients who have received antiviral medication including peramivir, laninamivir, oseltamivir, zanamivir, rimantadine, umifenovir, or amantadine within 7 days prior to the predose examinations
5. Patients who have received Chinese patent medicine or herbal medicine with antiviral effect within 7 days prior to the predose examinations
6. Patients who have received Anti-influenzal prescription within 7 days prior to the predose examinations
7. Subject who produces purulent sputum or has suppurative tonsillitis.
8. White blood cells(WBC)>10.0×109/L at screening.
9. Chest X - ray examination confirmed bronchitis,pneumonia,pleural effusion or pulmonary interstitial lesions.
10. Patients who have experienced respiratory tract infection,Otitis media,nasosinusitis.
11. Patients with severe or uncontrollable underlying diseases:blood disorders,severe chronic obstructive pulmonary disease(COPD),liver disorders(ALT or AST≥3 ULN,total bilirubin≥1.5 ULN),kidney disorders(serum creatinine>177μmol/L or 2mg/dL),chronic congestive heart failure(NYHA III-IV),mental disorders
12. Immunodeficiency,including malignant tumor,organ or marrow transplant,human immunodeficiency virus [HIV] infection,or patients receiving immunosuppressant therapy 3 months prior to enrollment.
13. Concomitant therapy with aspirin or salicylic acid.
14. Patients weighing < 40 kg or morbid obesity(Body mass index [BMI]≥30kg/m2)
15. Known history of alcohol abuse or drug abuse
16. Pregnancy or breastfeeding at screening and during the study.All female subjects of childbearing potential must have a negative urine pregnancy test at screening and during the trial.
17. Have received any other investigational products within 3 months prior to dosing.
18. Patients who, in the opinion of the investigator, would be unlikely to comply with required study visits, self-assessments, and interventions

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 750 (Actual)
Dates: Start 2020-12-28 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-05-16 (Actual)

PRIMARY OUTCOMES:
Time to Alleviation of Symptoms in Participants Randomized to ZSP1273 or Placebo | Up to 14 days after first dose
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of symptoms was defined as the time from the start of the study treatment to the time when all seven influenza-related symptoms were assessed by the participant as absent (0) or mild (1) for at least 21.5 hours.
  Time to alleviation of symptoms was analyzed using the Kaplan-Meier(KM) method; participants who did not experience alleviation of symptoms were censored at the last observation time point
Time to Alleviation of Symptoms in Participants Randomized to ZSP1273 or Oseltamivir | Up to 14 days after first dose
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of symptoms was defined as the time from the start of the study treatment to the time when all seven influenza-related symptoms were assessed by the participant as absent (0) or mild (1) for at least 21.5 hours.
  Time to alleviation of symptoms was analyzed using the Kaplan-Meier(KM) method; participants who did not experience alleviation of symptoms were censored at the last observation time point

SECONDARY OUTCOMES:
Percentage of Participants With Positive Influenza Virus Titer at Each Time Point in Participants Randomized to ZSP1273 or Placebo | Days 2, 4, 6
  Virus titer was quantified from nasopharyngeal swabs by tissue culture methods.
Percentage of Participants With Positive Influenza Virus Titer at Each Time Point in Participants Randomized to ZSP1273 or Oseltamivir | Days 2, 4, 6
  Virus titer was quantified from nasopharyngeal swabs by tissue culture methods.
Percentage of Participants With Positive Influenza Virus by RT-PCR at Each Time Point in Participants Randomized to ZSP1273 or Placebo | Days 2, 4, 6
  Influenza virus ribonucleic acid (RNA) was quantified from nasopharyngeal swabs.
Percentage of Participants With Positive Influenza Virus by RT-PCR at Each Time Point in Participants Randomized to ZSP1273 or Oseltamivir | Days 2, 4, 6
  Influenza virus ribonucleic acid (RNA) was quantified from nasopharyngeal swabs.
Change From Baseline in Virus Titer at Each Time Point in Participants Randomized to ZSP1273 or Placebo | Days 2, 4, 6
  Virus titer was quantified from nasopharyngeal swabs.
Change From Baseline in Virus Titer at Each Time Point in Participants Randomized to ZSP1273 or Oseltamivir | Days 2, 4, 6
  Virus titer was quantified from nasopharyngeal swabs.
Change From Baseline in Virus RNA (RT-PCR) at Each Time Point in Participants Randomized to ZSP1273 or Placebo | Days 2, 4, 6
  Nasopharyngeal swabs were obtained for viral quantitation.
Change From Baseline in Virus RNA (RT-PCR) at Each Time Point in Participants Randomized to ZSP1273 or Oseltamivir | Days 2, 4, 6
  Nasopharyngeal swabs were obtained for viral quantitation.
Area Under the Curve (AUC) Adjusted by Baseline in Influenza Virus Titer in Participants Randomized to ZSP1273 or Placebo | Up to 6 days after first dose
  This endpoint was defined as AUC of change from Baseline in virus titer from Day 1 to Day 5. AUC was calculated using the trapezoidal method
Area Under the Curve (AUC) Adjusted by Baseline in Influenza Virus Titer in Participants Randomized to ZSP1273 or Oseltamivir | Up to 6 days after first dose
  This endpoint was defined as AUC of change from Baseline in virus titer from Day 1 to Day 5. AUC was calculated using the trapezoidal method
Time to Cessation of Viral Shedding Determined by Virus Titer in Participants Randomized to ZSP-1273 or Placebo | Up to 6 days after first dose
Time to Cessation of Viral Shedding Determined by Virus Titer in Participants Randomized to ZSP1273 or Oseltamivir | Up to 6 days after first dose
Time to Cessation of Viral Shedding Determined by Virus RNA in Participants Randomized to ZSP1273 or Placebo | Up to 6 days after first dose
Time to Cessation of Viral Shedding Determined by Virus RNA in Participants Randomized to ZSP1273 or Oseltamivir | Up to 6 days after first dose
Percentage of Participants Whose Symptoms Were Alleviated at Each Time Point in Participants Randomized to ZSP1273 or Placebo | Up to 14 days after first dose
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms). Alleviation of symptoms was defined as all seven influenza-related symptoms assessed by the participant as absent (0) or mild (1)
Percentage of Participants Whose Symptoms Were Alleviated at Each Time Point in Participants Randomized to ZSP1273 or Oseltamivir | Up to 14 days after first dose
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms). Alleviation of symptoms was defined as all seven influenza-related symptoms assessed by the participant as absent (0) or mild (1)
Time to Alleviation of the Four Systemic Symptoms in Participants Randomized to ZSP1273 or Placebo | Up to 14 days after first dose
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of the 4 systemic symptoms was defined as the time between the initiation of the study treatment to the time when all 4 systemic symptoms (headache, feverishness or chills, muscle or joint pain, and fatigue) were assessed by the participant as 0 (None) or 1 (Mild) for a duration of at least 21.5 hours.
  Time to alleviation of the 4 systemic symptoms was analyzed using KM methods; participants who did not experience alleviation of symptoms were censored at the last observation time point.
Time to Alleviation of the Four Systemic Symptoms in Participants Randomized to ZSP1273 or Oseltamivir | Up to 14 days after first dose
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of the 4 systemic symptoms was defined as the time between the initiation of the study treatment to the time when all 4 systemic symptoms (headache, feverishness or chills, muscle or joint pain, and fatigue) were assessed by the participant as 0 (None) or 1 (Mild) for a duration of at least 21.5 hours.
  Time to alleviation of the 4 systemic symptoms was analyzed using KM methods; participants who did not experience alleviation of symptoms were censored at the last observation time point.
Time to Alleviation of the Three Respiratory Symptoms in Participants Randomized to ZSP1273 or Placebo | Up to 14 days after first dose
  * Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms). Time to alleviation of the 3 respiratory symptoms was defined as the time from the start of study treatment to the time when all 3 respiratory symptoms (cough, sore throat and nasal congestion) were assessed by the participant as absent (0) or mild (1) for at least 21.5 hours
  * Time to alleviation of the 3 respiratory symptoms was analyzed using the KM method; participants who did not experience alleviation of symptoms were censored at the last observation time point
Time to Alleviation of the Three Respiratory Symptoms in Participants Randomized to ZSP1273 or Oseltamivir | Up to 14 days after first dose
  * Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms). Time to alleviation of the 3 respiratory symptoms was defined as the time from the start of study treatment to the time when all 3 respiratory symptoms (cough, sore throat and nasal congestion) were assessed by the participant as absent (0) or mild (1) for at least 21.5 hours
  * Time to alleviation of the 3 respiratory symptoms was analyzed using the KM method; participants who did not experience alleviation of symptoms were censored at the last observation time point
Change From Baseline in Composite Symptom Score at Each Time Point in Participants Randomized to ZSP1273 or Placebo | Up to 14 days after first dose
  * Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms)
  * The composite symptom score is the total score of the 7 influenza symptoms as assessed by the participant at each time point
Change From Baseline in Composite Symptom Score at Each Time Point in Participants Randomized to ZSP1273 or Oseltamivir | Up to 14 days after first dose
  * Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms)
  * The composite symptom score is the total score of the 7 influenza symptoms as assessed by the participant at each time point
Time to Resolution of Fever in Participants Randomized to ZSP1273 or Placebo | Up to 14 days after first dose
  * Time to resolution of fever was defined as the time between the initiation of the study treatment and the resolution of fever. The resolution of fever was defined as the time when the participant's self-measured axillary temperature became less than 37ºC and was maintained at less than 37ºC for a duration of at least 12 hours
  * Time to resolution of fever was analyzed using KM methods; participants who did not experience resolution of fever by the last observation time point were censored at that time point
Time to Resolution of Fever in Participants Randomized to ZSP1273 or Oseltamivir | Up to 14 days after first dose
  * Time to resolution of fever was defined as the time between the initiation of the study treatment and the resolution of fever. The resolution of fever was defined as the time when the participant's self-measured axillary temperature became less than 37ºC and was maintained at less than 37ºC for a duration of at least 12 hours
  * Time to resolution of fever was analyzed using KM methods; participants who did not experience resolution of fever by the last observation time point were censored at that time point
Percentage of Participants Reporting Normal Temperature at Each Time Point in Participants Randomized to ZSP1273 or Placebo | Up to 14 days after first dose
  Defined as the percentage of patients whose axillary temperature dropped to less than 37ºC after the initiation of study treatment
Percentage of Participants Reporting Normal Temperature at Each Time Point in Participants Randomized to ZSP1273 or Oseltamivir | Up to 14 days after first dose
  Defined as the percentage of patients whose axillary temperature dropped to less than 37ºC after the initiation of study treatment
Time to Alleviation of Individual Symptoms in Participants Randomized to ZSP1273 or Placebo | Up to 14 days after first dose
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of each symptom was defined as the time from the start of treatment to the start of the time period when the individual symptom was assessed by the participant as 0 (None) or 1 (Mild) for a duration of at least 21.5 hours.
Time to Alleviation of Individual Symptoms in Participants Randomized to ZSP1273 or Oseltamivir | Up to 14 days after first dose
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Time to alleviation of each symptom was defined as the time from the start of treatment to the start of the time period when the individual symptom was assessed by the participant as 0 (None) or 1 (Mild) for a duration of at least 21.5 hours.
Time to Return to Preinfluenza Health Status in Participants Randomized to ZSP1273 or Placebo | Up to 14 days after first dose
Time to Return to Preinfluenza Health Status in Adults Randomized to ZSP1273 or Oseltamivir | Up to 14 days after first dose
  Defined as the time between the initiation of the study treatment and the return to normal activities of daily life. The return to normal activities of daily life is defined as the time when the subject assesses his/her activities as 10.Subjects with a baseline self-rated daily activity score of 10 are not included in this analysis.
Percentage of Participants With Influenza-related Complications in Participants Randomized to ZSP1273 or Placebo | Up to 14 days after first dose
  Defined as the time between the initiation of the study treatment and the return to normal activities of daily life. The return to normal activities of daily life is defined as the time when the subject assesses his/her activities as 10.Subjects with a baseline self-rated daily activity score of 10 are not included in this analysis.
Percentage of Participants With Influenza-related Complications in Participants Randomized to ZSP1273 or Oseltamivir | Up to 14 days after first dose
Change in EQ-5D-5L | Up to 14 days after first dose
  Defined as the change from baseline in the index value and that in EQ VAS score as calculated from the EQ-5D-5L questionnaire.

CONTACTS AND LOCATIONS:
Locations (76):
- China (76):
  - The First Affiliated Hospital of bengbu medical college, Bengbu, Anhui
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - Beijing Chaoyang Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Ditan Hospital Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - People's Hospital of Cuanjiang, Chongqing, Chongqing, Chongqing Municipality
  - Third Military Medical University, Chongqing, Chongqing Municipality
  - Quanzhou First Hospital, Quanzhou, Fujian
  - Fujian Provincal Hospital, Xiamen, Fujian
  - Xiamen Hospital of T.C.M, Xiamen, Fujian
  - Xiamen Zhongshan Hospital, Xiamen, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Foshan First People's Hospital, Foshan, Guangdong
  - Shunde University of Southern Medical University, Foshan, Guangdong
  - Guangdong Province Traditional Chinese Medical Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - Huizhou Central People's Hospital, Huizhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Qingyuan People's Hospital, Qingyuan, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - Yuebei People's Hospital, Shaoguan, Guangdong
  - Shenzhen Luohu Hospital Group Luohu People's Hospital, Shenzhen, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Songgang People's Hospital, Shenzhen, Guangdong
  - Nanning First People's Hospital, Nanning, Guangxi
  - Guizhou Provicial People's Hospital, Guiyang, Guizhou
  - Affiliated Hospital Zunyi Medical College, Zunyi, Guizhou
  - First Hospital of Qinhuangdao, Qinhuangdao, Hebei
  - Huaihe Hospital of Henan University, Huaihe, Henan
  - Luoyang Central Hospital Affiliated To Zhengzhou University, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Nanyang First People's Hospital, Nanyang, Henan
  - The Second People's hospital of Nanyang, Nanyang, Henan
  - The Third Affiliated Hospital of Nanyang Medical College, Nanyang, Henan
  - The Third Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Henan Provicial People's Hospital, Zhengzhou, Henan
  - Zhengzhou Central Hospital, Zhengzhou, Henan
  - Zhengzhou Sixth Hospital, Zhengzhou, Henan
  - Yiyang Central hospital, Yiyang, Hunan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Nanjing Jiangning Hospital, Nanjing, Jiangsu
  - Sir run run Hospital Nanjing Medical University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - First Affiliated Hospital of Gannan Medical University, Ganzhou, Jiangxi
  - Jiujiang University Affiliated Hospital, Jiujiang, Jiangxi
  - First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - The Third Hospital Of Nanchang, Nanchang, Jiangxi
  - Pingxiang People's Hospital, Pingxiang, Jiangxi
  - Shangyao People's Hospital, Shangyao, Jiangxi
  - The First Hospital Of Jilin University, Changchun, Jilin
  - General Hospital of Liaohe Oilfield, Panjin, Liaoning
  - Shenyang Central Hospital Affiliated To Shenyang medical college, Shenyang, Liaoning
  - Binzhou Medical University Hospital, Binzhou, Shandong
  - Heze Municipal Hospital, Heze, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - Linyi People's Hospital, Linyi, Shandong
  - Shandong Energy Zaozhuang Mining, Zaozhuang, Shandong
  - PKUCare luzhong Hospital, Zibo, Shandong
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - Chengdu Xinhua Hospital, Chengdu, Sichuan
  - General Hospital of Western Theater of PLA, Chengdu, Sichuan
  - Sichuan Provicial People's Hospital, Chengdu, Sichuan
  - The Third People's Hospital of Wuhou, Chengdu, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Dazhou Central Hospital, Dazhou, Sichuan
  - Affiliated Hospital of North Sichuan College, Nanchong, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The first People hospital of Yunnan Province, Kunming, Yunnan
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Ruian People's Hospital, Ruian, Zhejiang

REFERENCES:
- [Derived] Yang Z, Zhan Y, Li Z, Lin Z, Fang Z, Li H, Chen X, Ding B, Zeng H, Zhang X, Song Y, Lin Z, Liang S, Luo J, Huang J, Chen X, Zhong N; Onradivir Trial Recruitment and Medical Monitoring Group. Efficacy and safety of onradivir in adults with acute uncomplicated influenza A infection in China: a multicentre, double-blind, randomised, placebo-controlled and oseltamivir-controlled, phase 3 trial. Lancet Respir Med. 2025 Jul;13(7):597-610. doi: 10.1016/S2213-2600(25)00046-3. Epub 2025 Jun 7. PMID 40489986